CLINICAL TRIAL: NCT05562193
Title: Exercise Intervention Coupled With Standard Post-cancer Directed Treatment Care to Reduce Chronic Pain in Childhood Cancer Survivors Who Have Completed Cancer-directed Therapy Less Than One Year
Brief Title: Exercise and Pain in CCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Four Diamonds Research Fund at Penn State Health Childrens Hospital (Unknown)
Responsible Party: Principal Investigator, Smita Dandekar, Dr. Smita Dandekar, MD, Penn State Health Milton S Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00020762
Record Dates: First submitted 2022-09-26; First posted 2022-09-30 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Childhood Cancer Survivors

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical activity intervention coupled with standard post-cancer directed treatment care group (Experimental)
  Interventions: Behavioral: Physical activity intervention coupled with standard post-cancer directed treatment care
- Standard post-cancer directed treatment care control group (Other)
  Interventions: Other: Standard post-cancer directed treatment care control

INTERVENTIONS:
Behavioral: Physical activity intervention coupled with standard post-cancer directed treatment care — CCS will participate in a 16-week physical activity program. CCS will be instructed to start with a session duration of <15-min, three days per week at low intensity (e.g., activities expending >1.5 to 3 METs or intensity <5 on a scale of 0 to 10). Any type of physical activity will be acceptable. The program will be individualized, and activity increased according to patients' health status, results from the physical function assessment, and most recent week's achieved physical activities. The program will include support calls and texts from research staff (exercise physiologist). The program will be modified and adapted during support calls or texts, including frequency, intensity, time and type to maximize CCS' success. CCS will receive a Fitbit at the beginning of the intervention.
  Arms: Physical activity intervention coupled with standard post-cancer directed treatment care group
Other: Standard post-cancer directed treatment care control — CCS in the control group will not participate in a 16-week physical activity program and will not receive support calls or texts. Physical activity advice according to the Children's Oncology Group Guidelines for Diet and Physical Activity recommendations and the International Pediatric Oncology Exercise Guidelines will be offered to CCS following completion of 16-week follow-up. Moreover, CCS will receive a Fitbit following completion of 16-week follow-up
  Arms: Standard post-cancer directed treatment care control group

SUMMARY:
The purpose of this study is to demonstrate that integration of exercise intervention into standard post-cancer directed treatment care will improve patient reported pain, decrease the need for medications to manage chronic pain and improve functional and psychosocial outcomes in survivors of cancers in children and adolescents. Our central hypothesis is that integration of exercise interventions into standard post-cancer directed treatment care will be acceptable and feasible while improving patients' pain, decreasing the cumulative dose of pain medication and improving patients' functional and psychosocial outcomes as compared to patients who only receive standard post-cancer directed treatment care.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female CCS diagnosed with any type of cancer
2. CCS who have completed all standard/planned cancer treatment and are stable at the time of recruitment
3. CCS are < 1-year post cancer therapy
4. CCS who have chronic pain (pain will be self-reported by the participant, will have to be ≥1 on a scale of 10 and lasting for 3 months or longer)
5. CCS who are age between 10 and 17 years old at the time of enrollment
6. CCS who are and who are not non-ambulatory/wheelchair bound.
7. CCS and parent/legal guardian must be able to speak, read and understand the English language
8. CCS's parent or legal guardian must be able to provide and understand informed consent
9. CCS must be able to provide and understand assent
10. CCS must be able to attend three visits (baseline, 8 and 16-week follow-up) at the Penn State Health Children's Hospital
11. CCS and parent/legal guardian must have access to a computer, smartphone or tablet

Note: The agreement of the attending oncologist will be required for the participation of CCS eligible for this study.

Exclusion Criteria:

1. CCS who have not completed all standard/planned cancer treatment and/or not in complete remission at the time of recruitment
2. CCS who are > 1-year post cancer therapy
3. CCS who are < 10 years old and > 17 years old at the time of enrollment
4. CCS who have evidence in their medical record of an absolute contraindication to complete any of the physical assessments in their medical record. This exclusion criterion is at the oncologist's discretion when research staff will contact the medical oncologist via secure email or secure message through the electronic medical record for approval to approach their patients for the study and for medical clearance. The oncologists can update this information at any time during the study if there is evidence of an absolute contraindication to complete any of the physical assessments.
5. CCS who have history of refractory or recurrent cancer
6. CCS or their parent/legal guardian who are unable to speak, read, and understand the English language
7. CCS who are unable to access and complete online questionnaires

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
Acceptability of the intervention | Baseline
  The number of participants approached who agree to participate in the study
Feasibility of the intervention | Baseline to week 16
  The number of participants randomized to the physical activity program intervention coupled with standard post-cancer directed treatment care who complete at least 50% of the physical activity intervention.

SECONDARY OUTCOMES:
Measure changes in chronic pain levels | Baseline, week 8 and week 16
  Self-reported chronic pain questionnaire using the PedsQL pediatric pain questionnaire. The parent proxy-report format is used to assess the parent's perceptions of their child's pain.
  Range 0-100, Higher score indicates higher pain intensity
Measure changes in cumulative dose of pain medications | Baseline, week 4, week 8, week 12 and week 16
  * Chart review: number of pain medications prescribed, total dosage and length of time prescribed.
  * Self-reported pain medication: usage of prescription medication and information about the use of non-prescription pain medications (e.g., over the counter oral and topical pain medications).
  * The Prescription Drug Monitoring Program will be accessed to gather information on all filled prescriptions for controlled substances within the state of Pennsylvania.
  * Morphine equivalent dose will be calculated for each patient after looking at the total daily amount of each opioid the patient is taking. Using the standard conversion factors developed by the CDC, the Morphine milligram equivalent equates the many different opioids into a standard value that is based on morphine and its potency providing an easily interpretable metric for representing opioid utilization
Measure changes in patient reported outcomes | Baseline, week 8 and week 16
  Psychosocial questionnaires using the NIH developed PROMIS pediatric questionnaires, which are validated for pediatric oncology, including: Self-reported physical function mobility, Anxiety, Depressive symptoms, Fatigue, Peer relationships, Social isolation, Pain interference, Pain intensity, Sleep disturbance, Cognitive function.
  PROMIS pediatric questionnaires assessing PROs on 5 point Likert scale responses
Measure changes in physical activity level | Baseline, week 8 and week 16
  Self-reported physical activity questionnaire using the Godin-Shephard leisure-time physical activity questionnaire.
  * Less than 14 units: Insufficiently active
  * 14 to 23 units: Moderately active
  * 24 units or more: Active
Measure changes in patient functional outcomes (6-min walking test) | Baseline and week 16
  Validated physical function tests for pediatric patients, including the 6-min walking test Further distances indicate greater physical function
Measure changes in patient functional outcomes (30-second chair stand test) | Baseline and week 16
  Validated physical function tests for pediatric patients, including the 30-second chair stand test Greater amounts of sit/stands indicate greater physical function
Measure changes in patient functional outcomes ("Timed Up and Go" test) | Baseline and week 16
  Validated physical function tests for pediatric patients, including the "Timed Up and Go" test Shorter durations indicate greater physical function
Measure changes in patient functional outcomes (grip strength test) | Baseline and week 16
  Validated physical function tests for pediatric patients, including the grip strength test Greater grip strength indicate greater physical function

CONTACTS AND LOCATIONS:
Overall Officials: Smita Dandekar, MD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Health Children's Hospital, Hershey, Pennsylvania, United States